CLINICAL TRIAL: NCT01803685
Title: A Nationwide Treatment Survey of Intracranial Arteriovenous Malformation: a Multicenter Retrospective and Prospective Register Study in China
Brief Title: Nationwide Treatment Survey of Intracranial Arteriovenous Malformation in China
Acronym: NTSIAVMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Yong Cao (Other)
Responsible Party: Sponsor-Investigator, Dr. Yong Cao, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: IAVM-125R
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Intracranial Arteriovenous Malformations
Keywords: Intracranial Arteriovenous Malformations; Surgical removal; Endovascular embolism; Stereotaxic radiosurgery; Outcomes
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Surgical treatment: Surgical resection of intracranial arteriovenous malformations.
- Stereotaxic radiosurgery: Deliver a relatively high dose of focused radiation precisely to the arteriovenous malformations.
- Endovascular treatment: Deliver embolic materials to the feeding arteries or the nidus by microcatheters
- Comprehensive treatment: Use two or three methods ( Surgical treatment stereotaxic radiosurgery endovascular treatment ) to cure the intracranial arteriovenous malformations
- Conservative treatment: Patients refused to any of the treatment above

SUMMARY:
This register study will collect the treatment information of the intracranial arteriovenous malformation patients in China. We aim to understand the current treatment situation of the disease in China.

DETAILED DESCRIPTION:
Intracranial arteriovenous malformations are congenital lesions that consist of multiple arteries and veins, connecting as a fistula without intervening normal capillary bed. The treatment strategy including surgical removal, endovascular embolism and stereotaxic radiosurgery and comprehensive treatment. China is a united multi-ethnic nation of 56 ethnic groups, and has the largest population in the world. We have most extensive and valuable clinical resources of intracranial arteriovenous malformation in the world. But we know little about the current treatment situation of the disease in China.

In order to realize the treatment situation of intracranial arteriovenous malformation in China, we designed a retrospective and prospective register study to collect the treatment and outcome information all over China.

ELIGIBILITY:
Inclusion Criteria:

* All the patients that diagnosed of intracranial AVM by DSA/CT/MRI
* All patients gave written informed consent

Exclusion Criteria:

* patients refuse to attend the survey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients that diagnosed of intracranial AVM by DSA/CT/MRI
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
modified Ranking Scale | six months after operation
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead

SECONDARY OUTCOMES:
Treatment complications | six months after treatment
  Post operative epilepsy seizure, hemorrhage,infarction;cerebral edema、endovascular embolization injury

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Department of Neurosurgery, Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China